CLINICAL TRIAL: NCT01271595
Title: Acupuncture in Seasonal Allergic Rhinitis- Effects on the Autonomic Nervous System (AUTO-ACUSAR)- an Explorative Substudy of ACUSAR
Brief Title: AUTO-ACUSAR - Effects of Acupuncture on the Autonomic Nervous System in Seasonal Allergic Rhinitis Patients
Acronym: AUTO-ACUSAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Prof. Dr. Benno Brinkhaus, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EA1/214/07a
Record Dates: First submitted 2010-12-23; First posted 2011-01-07 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: acupuncture; autonomic nervous system; seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture (Active Comparator): 12 sessions of acupuncture according to TCM
  Interventions: Other: sham acupuncture
- sham acupuncture (Sham Comparator): superficial acupuncture at non acupuncture sites
  Interventions: Other: sham acupuncture

INTERVENTIONS:
Other: sham acupuncture — 12 sessions of sham acupuncture over 8 weeks
  Other Names: acupuncture

SUMMARY:
There is inconclusive evidence whether acupuncture treatment is effective in the treatment of seasonal allergic rhinitis (SAR). Furthermore, the underlying mechanisms of acupuncture in SAR are only poorly understood. It was hypothesised that the therapeutic mechanism of acupuncture is related to changes in autonomic function. AUTO-ACUSAR is a sub-study of the DFG-funded three-arm randomized controlled trial ACUSAR trial investigating the efficacy of acupuncture vs. sham acupuncture vs. rescue medication in SAR. The aim of AUTO-ACUSAR was to investigate short and long-term effects of acupuncture vs. sham acupuncture on autonomic function in a sub-group of ACUSAR patients. Baseline values were compared to data from matched healthy controls.

DETAILED DESCRIPTION:
In AUTO-ACUSAR a subsample of ACUSAR patients from acupuncture or sham acupuncture groups were included. Tests of autonomic functions included measurement of heart rate variability during paced breathing, blood pressure, heart rate and salivary alpha amylase response to a cold pressure test (CPT) and cortisol awakening response before the first and the last of twelve treatment sessions. Healthy matched controls underwent the same measurement once only

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients (aged 16-45 years) with seasonal allergic rhinitis, clinically positive and test positive (skin-prick test and/or RAST) to grass and birch pollen
* Patients with >2 years of moderate to severe SAR
* Positive skin-prick test and/or RAST (at least class 2) results
* Visual analogue scale >40mm and <80 mm for SAR symptoms during the past year
* Patients must be able to complete a diary for self-evaluation of symptoms and recording use of anti-symptomatic medication
* Use of, or indication for, oral antihistamines as anti-allergic medication
* Written informed consent

Exclusion Criteria:

* Perennial SAR or other types of chronic rhinitis
* Allergic asthma and/or moderate to severe atopic dermatitis
* Active tuberculosis
* Auto-immune disorders
* Severe chronic inflammatory diseases
* History of anaphylactic reactions
* Hypersensitivity to Rescue medication or related drugs used in study related drugs
* Specific immunotherapy >3 years
* Simultaneous participation in other clinical trials
* Serious acute or chronic organic disease or mental disorder
* Pregnancy or breast feeding
* Allergy desensitisation therapy (current, during the past two years, or planned in the next two years)
* Blood coagulation disorder and/or current use of anticoagulants
* Previous acupuncture treatment for SAR
* Any Complementary and alternative medicine treatment at the moment, in the last three months or planned in the next two years

  * intake of Beta-Blocker Medication
  * use of pacemaker

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 8 weeks
  RMSSD, LF, HF, HR, blood pressure

SECONDARY OUTCOMES:
Salivary Amylase and Cortisol, Cortisol Awakening Response (CAR) | 8 weeks
  Measurements were taken during the experimental setting 3 times , CAR by the patients the day before first and last acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Benno Brinkhaus, Prof. Dr., Principal Investigator — Institute for Socialmedicine, Epidemiology and Health Economics, Charité University Medical Center
Locations (1):
- Institute for Socialmedicine, Epidemiology and Health Economics, Charité University Medical Center, Berlin, Germany